CLINICAL TRIAL: NCT00913861
Title: Does Non-pharmacological Intervention Reduce Consumption of Propofol During Colonoscopy?
Brief Title: Non-pharmacological Intervention for Colonoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: affiliation's change of the principal investigator need a new review bord
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Cheseaux Nicole, MD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-238; NAC 08-072
Record Dates: First submitted 2009-05-22; First posted 2009-06-04 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Colonoscopy; Sedation; Hypnosis
Keywords: endoscopy; comfort; non-pharmacological
MeSH Terms: interventions — Hypnosis; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- standard sedation (Active Comparator): propofol and fentanyl
  Interventions: Drug: standard sedation
- structured attention-standard sedation (Active Comparator): structured attention
  Interventions: Behavioral: Structured attention
- hypnosis-standard sedation (Experimental): hypnosis
  Interventions: Behavioral: hypnosis

INTERVENTIONS:
Behavioral: hypnosis — Hypnosis: induction of hypnosis by visual fixation and recollection of a pleasant memory, suggestion of relaxation, of self-control and post-hypnotic suggestion for bowel relaxation.
  Other Names: hypnotic state
  Arms: hypnosis-standard sedation
Drug: standard sedation — Standard sedation: fentanyl 2x0,5 microg/kg at beginning of procedure and propofol PCS: 20mg bolus than 10mg/bolus, lock-out = 0.
  Other Names: Disoprivan (propofol)and fentanyl
  Arms: standard sedation
Behavioral: Structured attention — Structured attention: verbal and nonverbal communication; attentive listening; provision of the perception of control; encouragement; use of emotionally neutral descriptors, focus on a sensations.
  Other Names: psychological support
  Arms: structured attention-standard sedation

SUMMARY:
The purpose of this study is to determine whether a non-pharmacological intervention reduces consumption of sedative drugs during colonoscopy. A reduction of sedative drugs may reduce side effects. This non-pharmacological intervention may increase patient's comfort and security.

DETAILED DESCRIPTION:
Sedative and analgesic drugs are used in most patients related to pain and anxiety during the colonoscopy. Analgesia and sedation has adverse effects such as central respiratory depression, obstruction of the upper airways, hypoxia, hypotension and bradycardia. Non-pharmacological interventions had beneficial effects during percutaneous vascular or renal procedures. In this study we test the hypothesis that the adjunction of hypnosis to pharmacological sedation will decrease the quantity of sedative drugs used and will reduce the patient's anxiety and discomfort.

ELIGIBILITY:
Inclusion Criteria:

* patients classified as ASA 1 to 3
* colonoscopy with anesthesiological support
* capacity of consenting

Exclusion Criteria:

* pregnancy
* colonoscopy with gastroscopy
* emergency
* psychotic diseases
* deafness
* incapacity to understand french
* addiction of drugs and alcohol
* psychoactive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
total dose of propofol | the day of the colonoscopy, at the end

SECONDARY OUTCOMES:
gastroenterologist's satisfaction and quality of the colonoscopy | the day of the procedure, at the end of the procedure
vital parameters | during all the procedure, every 5 minutes
patient's comfort | during the procedure every 10 minutes and 1 and 14 days after the colonoscopy
anxiety state | between 30 minutes to one hour before coloscopy and between 5 minutes and 1 hour after the end of the procedure
patient's satisfaction | between 5 minutes to 1 hour after the end of the procedure and 1 and 14 days after the colonoscopy
duration of the procedure | the day of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Cheseaux, MD, Principal Investigator — Division of Anesthesiology, University Hospitals, Geneva
Locations (1):
- Division of Anesthesiology, University Hospitals of Geneva, Geneva, Canton of Geneva, Switzerland